CLINICAL TRIAL: NCT01271270
Title: A Phase I Unmasked Study to Investigate the Safety and Tolerability of Subconjunctival Injections of Palomid 529 in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Palomid 529 in Patients With Neovascular Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110066; 11-EI-0066
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2012-09-20

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-Related Macular Degeneration (AMD); Palomid 529; Age Related Macular Degeneration; AMD
MeSH Terms: conditions — Macular Degeneration | interventions — palomid 529

INTERVENTIONS:
Drug: Palomid 529

SUMMARY:
Background:

* Wet age-related macular degeneration (AMD) occurs when abnormal blood vessels grow in the back of the eye, and leak blood and other fluids that damage the eye, produce scarring, and lead to blindness. People diagnosed with wet AMD have increased production of a body chemical called vascular endothelial growth factor (VEGF). VEGF is important in the formation of blood vessels in the body, and decreasing the production of VEGF is believed to help wet AMD patients by preventing or slowing the growth of the abnormal blood vessels. Anti-VEGF drugs have been used to decrease the production of VEGF, but some people do not respond completely to these drugs.
* A protein in the body called mTOR also plays a critical role in regulating how cells divide and grow and obtain their blood supply. The experimental chemical Palomid 529 inhibits the production of mTOR. Researchers are interested in determining whether Palomid 529 is safe and can help individuals with wet AMD who have not completely responded to anti-VEGF treatments.

Objectives:

- To evaluate the safety and effectiveness of Palomid 529 as a treatment for wet age-related macular degeneration in individuals who have not responded to standard anti-VEGF treatments.

Eligibility:

- Individuals with wet age-related macular degeneration in at least one eye that has not responded to standard anti-VEGF treatments.

Design:

* Prior to the first visit, participants should have been seen at the National Eye Institute clinic under a screening or teaching protocol, or NIH protocol 08-EI-0103, High Speed Indocyanine Green Angiography Findings in Induction Regimen of Intravitreal Ranibizumab Injection for Neovascular Age Related Macular Degeneration. One eye will be designated as the study eye to receive the Palomid 529 treatment.
* Participants will have a full physical examination and medical history, a full eye examination to evaluate eye health and vision, angiography to examine the blood vessels in the eyes, and blood and urine tests during the study
* Participants will receive an injection of Palomid 529 into the study eye every 4 weeks during the study, for a total of three injections. Participants may also receive anti-VEGF injections such as ranibizumab (Lucentis ) or bevacizumab (Avastin ) in the study eye 12 days before and 12 days after the Palomid 529 injection.
* Participants may have standard-of-care treatments for the non-study eye if it has wet AMD as well, but may not receive experimental treatments in the non-study eye while they are in this study.
* Participants will return for long-term follow-up examinations as directed by the study researchers.

DETAILED DESCRIPTION:
Objective:

Paloma Pharmaceuticals, Inc. has developed a non-steroidal, wholly synthetic, small molecule drug for application to diseases of aberrant neovasculature, known as Palomid 529.1 Palomid 529 exerts broad activity as an anti-angiogenic agent by inhibiting the mammalian target of rapamycin (Akt/mTor) signal transduction pathway via dissociation of both target of rapamycin complexes (TORC1 and TORC2) in the immune system.

The objective of this study is to evaluate the safety and tolerability of Palomid 529 when administered as subconjunctival injections in participants with choroidal neovascularization (CNV) secondary to neovascular age-related macular degeneration (AMD).

Study Population:

This study will enroll participants with neovascular AMD who have not responded to conventional anti-VEGF treatments. Five participants will be initially accrued; however, up to seven participants who meet the eligibility criteria may be enrolled.

Design:

This is a 12-week, unmasked, non-randomized study of three serial 1.9 mg subconjunctival doses of Palomid 529 in neovascular AMD participants who have not responded to conventional anti-VEGF treatments.

Outcome Measures:

The primary outcome is to determine the safety of subconjunctival Palomid 529 for neovascular AMD. Safety outcomes include the number and severity of ocular and systemic adverse events. Secondary efficacy outcomes include changes in best-corrected visual acuity (BCVA), changes in fluid status, central retinal thickness and retinal volume as measured by optical coherence tomography (OCT), changes in leakage patterns as observed on fluorescein angiography (FA), changes in CNV patterns as observed on indocyanine green angiography (ICG), changes in autofluorescence patterns as observed on fundus autofluorescence (FAF) imaging, and changes in fundus appearance as observed on color fundus photography. Additionally, Complement Factor H polymorphisms will be compared with treatment response and pharmacokinetic samples will be collected.

ELIGIBILITY:
* STUDY EYE INCLUSION CRITERIA:

  1. Participant must have active neovascular AMD in at least one eye (the study eye) as defined by the following criteria:

     * CNV in the setting of AMD resulting in fluid or blood within the macula as determined by clinical examination, OCT or FA.
     * The study eye has not responded to conventional anti-VEGF treatment (defined as the eye that has any persistent intraretinal cyst with a greatest linear dimension of at least 100 microns and/or subretinal fluid pocket with a height of at least 100 microns and/or the presence of any foveal fluid after four serial anti-VEGF intravitreal injections). The fluid state will be determined two weeks (plus or minus two days) after the last injection.
  2. Participant must have reasonably clear media and some fixation to allow for good quality OCT and fundus photography.
  3. Participant must have visual acuity of 20 over 40 or worse in the study eye. Participants who meet all other eligibility criteria and have visual acuity between 20 over 32 and 20 over 40 may be enrolled if their disease is considered vision-threatening as determined by the investigator (i.e., they have persistent fluid under the fovea and are not responding to standard-of-care anti-VEGF treatment).

INCLUSION CRITERIA:

* Participant must be 18 years of age or older.
* Participant must understand and sign the protocol s informed consent document.
* Female participants of childbearing potential must not be pregnant or lactating, must have a negative pregnancy test at screening and must be willing to undergo pregnancy tests throughout the study.
* Women of childbearing potential must agree to use reliable methods of contraception during the study period and for three months following the last injection. Acceptable methods of contraception include hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom with spermicide) or surgical sterilization (hysterectomy, tubal ligation or partner with vasectomy).

EXCLUSION CRITERIA:

* Participant is actively receiving another investigational study therapy. Participation in NIH protocol 08-EI-0103, High Speed Indocyanine Green Angiography Findings in Induction Regimen of Intravitreal Ranibizumab Injection for Neovascular Age-Related Macular Degeneration is allowed, if s/he has been enrolled for at least one year, as this is an imaging study providing standard-of-care ranibizumab.
* Participant is unable to comply with study procedures or follow-up visits.
* Participant has evidence of ocular disease other than neovascular AMD in the study eye that may confound the outcome of the study (i.e., diabetic macular edema, myopic choroidal neovascularization or uveitic macular edema).
* Participant has evidence of retinal pigment epithelial detachment (unless subretinal or intraretinal fluid is present)in the study eye.
* Participant received an anti-VEGF injection in the study eye within 12 days prior to enrollment.
* Participant received or has been receiving intraocular steroids in the study eye within four months prior to enrollment.
* Participant received or has been receiving immunosuppressive treatments (i.e., biologic or systemic steroids) within two months prior to enrollment. If the participant was on any systemic immunosuppressive treatment for at least two months prior to enrollment and meets the enrollment criteria of residual fluid after four serial anti-VEGF injections, then s/he is eligible to participate in the study as long as s/he will continue this specific systemic drug regimen for the entire study period.
* Participant is allergic to fluorescein dye or indocyanine green dye.
* Participant is allergic to shellfish or iodine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-12-20; Primary Completion 2012-09-20 (Actual); Study Completion 2012-09-20 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to determine the safety of subconjunctival Palomid 539 neovascular AMD. Safety outcomes include the number and severity of ocular and systemic adverse events.

SECONDARY OUTCOMES:
Efficacy outcomes include changes in BCVA, fluid status, central retinal thickness, retinal volume, leakage patterns, CNV patterns and fundus appearance. Collecting Complement Factor H Genotypes and pharmacokinetic samples.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Meyerle, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Dalal M, Jacobs-El N, Nicholson B, Tuo J, Chew E, Chan CC, Nussenblatt R, Ferris F, Meyerle C. Subconjunctival Palomid 529 in the treatment of neovascular age-related macular degeneration. Graefes Arch Clin Exp Ophthalmol. 2013 Dec;251(12):2705-9. doi: 10.1007/s00417-013-2375-7. Epub 2013 May 21. PMID 23689994